CLINICAL TRIAL: NCT06091319
Title: Florbetaben for Imaging of Vascular Amyloid: Evaluation of Amyloid Inflammasome Imaging in Carotid and Coronary Arteries in Patients With Unstable Atherosclerosis- A Pilot Study
Brief Title: Florbetaben for Imaging of Vascular Amyloid
Acronym: FERMATA
Status: Recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 1.0
Record Dates: First submitted 2023-08-11; First posted 2023-10-19 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Acute Coronary Syndrome; Stroke; Transient Ischemic Attack; Atherosclerosis of Artery
MeSH Terms: conditions — Acute Coronary Syndrome; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute atherosclerotic disease event group: Patients with a recent ACS (i.e. STEMI or NSTEMI), stroke or transient ischemic attack.
- Control: A control population of patients with known vascular disease but without recent ACS, stroke/TIA.

SUMMARY:
The Primary Objective is to determine if a new nuclear tracer (named 18F-Florbetaben) used with nuclear imaging (PET imaging) can detect inflamed plaque in patients with recent ACS or stroke/TIA.

DETAILED DESCRIPTION:
The Primary Objective is to determine the feasibility of using 18F-Florbetaben PET in patients with recent ACS or stroke/TIA to detect inflammatory plaque.

Exploratory Objectives will define relationships of calcification imaging to other biomarkers and comparisons between high and low plaque burden regions and between patients with and without recent vascular events.

Patients with a recent ACS (i.e. STEMI or NSTEMI), stroke or transient ischemic attack (TIA) will be recruited will be recruited to the FERMATA study. A control population of patients with known vascular disease but without recent ACS, stroke/TIA will also be recruited.

FERMATA is a pilot, single- centerre, imaging study. We will evaluate the ability of the amyloid tracer, 18F-Florbetaben, to detect active atherosclerotic plaque in patients with recent ACS, or recent TIA/stroke. We plan to enroll 24 patients with ACS or patients with stroke/TIA and 6 control patients without recent ACS or stroke/TIA. Primary endpoint is the difference in Florbetaben uptake between the culprit artery (of either the ACS or TIA/stroke, respectively), and the non-culprit arteries. Parameters of interest are the maximal and total standard uptake values (SUVs) and tissue-to- background ratios (TBRs) of the coronary and carotid arteries as well as aorta.

Exploratory endpoints include a correlation analysis (Pearson correlation) to evaluate the relationship of inflammation on Florbetaben PET/CT to the histopathological levels of inflammation. In addition, we will look to see if Florbetaben uptake on PET correlates with lesion levels of B-amyloid. Comparisons will also be made between regions of high plaque burden vs lower plaque burden and between patients with recent vascular events vs those who have not had recent events.

ELIGIBILITY:
Inclusion Criteria:

1. suffered a recent cardiovascular event (30-120 days post ACS (i.e. STEMI or NSTEMI) or TIA/stroke with ipsilateral large vessel atherosclerotic disease confirmed on US, CT or MRI;
2. stable symptoms and hemodynamics;
3. age >/= 18 years;
4. given informed consent.

Exclusion Criteria:

1. a recent CV event likely to have been embolic in the opinion of the neurologist or cardiologist;
2. severe LV dysfunction (EF<30%);
3. severe valve disease requiring intervention;
4. decompensated heart failure;
5. pregnancy (all women of child bearing potential will have a negative BHCG test;
6. breastfeeding;
7. women of childbearing potential who refuse to use two forms of contraception (this includes at least one form of highly effective and one effective method of contraception) throughout the study OR men capable of fathering a child who refuse to use contraception;.
8. unable to give informed consent;.
9. Florbetaben allergy;
10. glomerular filtration rate (GFR) <50 ml/min/1.72m2

Exclusion for CTA portion of the protocol: Patients with dye allergy, or those with GFR <60, will not undergo CTA but will have PET/CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a recent ACS (i.e. STEMI or NSTEMI), stroke or transient ischemic attack (TIA) will be recruited. Standard definitions will be used for STEMI, NSTEMI including chest pain, EKG changes and troponin rise; likewise for ischemic stroke confirmed by CT or MRI imaging and TIA confirmed as a definite by a neurologist.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using 18F-Florbetaben PET in patients with recent ACS or stroke/TIA to detect inflammatory plaque | Within 16 weeks of vascular event
  Ratio of the standardized uptake value (SUV) of Florbetaben tracer to the background (SVC or internal jugular for coronary or carotid respectively)

OTHER OUTCOMES:
TBR of arteries in acute patients compared to control patients | Within 16 weeks of vascular event
  Tissue to background (TBR) of arteries in patients with acute vascular events compared to TBR in arteries of control patients
TBR of arteries in with higher plaque burden compared to lower plaque burden | Within 16 weeks of vascular event
  Tissue to background (TBR) of arteries in patients with higher plaque burden on CT compared to TBR in arteries of lower plaque burden

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Boczar, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided